Principal Investigator: Michael Goldfarb, PhD. Version Date: February 4, 2016

Study Title: Mobility and therapeutic benefits resulting from exoskeleton use in a clinical setting (SC140121 Study 1).

Institution/Hospital: Vanderbilt University and Medical Center

## **Statistical Analysis Plan**

## Mobility and Therapeutic Benefits resulting from Exoskeleton Use in a Clinical Setting (SC140121 Study 1)

## NCT03082898

Michael Goldfarb, PhD
H. Fort Flowers Professor of Mechanical Engineering
Professor of Electrical Engineering
Professor of Physical Medicine and Rehabilitation
VU Station B351592
2301 Vanderbilt Place
Nashville TN 37235

## Statistical Analysis Plan

Normality of data was determined for each measure by a Kolmogorov–Smirnov (KS) test. All measures were determined to be non-normally distributed, and as such are represented by median and IQR rather than mean and standard deviation. Differences in medians in all measures were tested using a Wilcoxon rank-sum test, with confidence levels for each given by corresponding p values.